CLINICAL TRIAL: NCT03912558
Title: Prospective, Open-Label, Non-Comparative, Pilot Study to Assess the Safety and Efficacy of Butterfly Medical Prostatic Retraction Device in Benign Prostatic Hyperplasia (BPH) Patients.
Brief Title: Pilot Study to Assess the Safety and Efficacy of Butterfly Medical Prostatic Retraction Device in BPH Patients.
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Butterfly Medical Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: BM-011
Record Dates: First submitted 2019-04-07; First posted 2019-04-11 (Actual); Last update posted 2024-08-06 (Actual); Status verified 2024-08

CONDITIONS: BPH; BOO - Bladder Outflow Obstruction
Keywords: BPH; BOO; Enlarged prostate; LUTS; Urinary obstruction; Retrograde ejaculation
MeSH Terms: conditions — Retrograde Ejaculation

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Butterfly device implantation (Experimental): Butterfly device implantation will be performed following initial cystoscopy to evaluate prostate condition and rule out other pathologies.
  Following implant size selection, the Butterfly implant will be deployed and positioned through the cystoscope over-sheath. After deployment the cystoscope (with its optics) will be re-introduced into the urethra to examine the Butterfly device position.
  Interventions: Procedure: Butterfly device implantation

INTERVENTIONS:
Procedure: Butterfly device implantation — The Butterfly device will be positioned and deployed with cystoscopy guidance

SUMMARY:
This study evaluates the safety and efficacy of use of the Butterfly Medical's prostatic retraction device in Benign Prostatic Hyperplasia (BPH) Patients. The study follows patients implanted with the Butterfly device for up to 1 year after implantation.

Evaluations include recording of safety events and BPH related symptoms by Uroflowmetry tests and International Prostate Symptom Score (IPSS) questionnaires. The study also assess sexual quality of life after implantation of the Butterfly device.

DETAILED DESCRIPTION:
Benign prostatic hyperplasia (BPH) is a non-cancerous enlargement of the prostate gland that may restrict the flow of urine from the bladder. BPH is a cellular proliferative process of the prostate, also referred as enlarged prostate.

An estimated 50% of men demonstrate histopathologic BPH by age 60 years. This number increases to 90% by age 85 years; thus, increasing gland size is considered a normal part of the aging process.

Approximately half of those diagnosed with histopathologic BPH demonstrate moderate-to-severe BPH related symptoms (also known as Lower Urinary Tract Symptoms = LUTS), including urinary frequency, urgency, nocturia (getting up at night during sleep to urinate), decreased or intermittent force of stream, or a sensation of incomplete emptying. Complications occur less commonly but may include acute urinary retention, impaired bladder emptying, or the need for surgery.

In current clinical practice, most patients are initially treated with medical therapy, usually with alpha-blockers. A minimally invasive treatment alternative is the use of urethral stents to preserve flow of urine from the bladder. Such stents are also associated with several problems such as encrustation, stone formation, pain, infection, migration and others. Another alternative is the gold standard treatment for managing benign prostatic hyperplasia; the trans urethral resection of prostate (TURP) surgery. Complications associate with TURP procedure include retrograde ejaculation, urinary incontinence, erectile dysfunction, urethral stricture, and others.

The Butterfly Medical Prostatic Retraction Device is a definitive device intended for transurethral insertion into the male prostatic urethra diagnosed with Bladder Outlet Obstruction (BOO), caused by an enlarged prostate gland. It is a single use device intended to remain permanently in the prostate urethra, to open the occluded urethral passage. The Butterfly device has a specific shape adjusted to fit the prostatic urethral lumen, and is designed to reside only in the prostate urethra without migration to the urinary bladder or the bulbar urethra. Unlike other forms of treatment, the Butterfly device does not inflict any damage to the bladder neck, preventing irritation or retrograde ejaculation.

ELIGIBILITY:
Inclusion Criteria:

1. Age 50 or older
2. Verified BPH with prostate size of at least 30 grams or of 25 mm.
3. Signed Informed Consent
4. Failure, intolerance or patient non-compliance of medical treatment
5. Patients suffering from LUTS symptoms of BPH (IPSS >12, Qmax=<13 ml/sec)
6. Patient's voided volume of at least 125 ml in uroflow test
7. Patients not eligible for surgery or refusing surgery

Exclusion Criteria:

1. Known sensitivity to Nickel
2. Active Prostatitis
3. Urethral strictures
4. Prior surgery of prostate (simple or radical)
5. Currently active bladder tumor
6. Suspected neurogenic urinary bladder
7. Suspected a-contractile bladder
8. Enlarged median lobe of prostate.
9. Bladder Neck stricture or contracture
10. Urethral pathology: diverticula, strictures, tumors, fistula
11. Clinically Significant urinary tract infection
12. Uncontrolled bleeding disorders
13. Uncontrolled diabetes mellitus
14. Severe medical diseases precluding a minimally invasive procedure
15. Present active urinary stone disease
16. Patients who are under anticoagulants therapy

Min Age: 50 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 92 (Actual)
Dates: Start 2018-10-29 (Actual); Primary Completion 2024-04-01 (Actual); Study Completion 2024-04-01 (Actual)

PRIMARY OUTCOMES:
Reported device related adverse events | 12 months post procedure
  Assess the rate, nature and severity of device-related adverse events reported
Cystoscopic assessment - inflammation | 12 months post procedure
  Cystoscopic assessment to evaluate lack of local inflammation
Cystoscopic assessment - incrustations | 12 months post procedure
  Cystoscopic assessment to evaluate no incrustations
Cystoscopic assessment - implant coverage | 12 months post procedure
  Cystoscopic assessment to evaluate coverage by mucosa
Device migration | 12 months post procedure
  Rate of migration of the Butterfly device

SECONDARY OUTCOMES:
Symptoms reduction - IPSS | Baseline to 12 months post procedure
  Improvement in IPSS at 12 months compared to baseline
Symptoms reduction - Qmax | Baseline to 12 months post procedure
  Improvement in Qmax (by uroflowmetry) at 12 months compared to baseline
Sexual quality of life evaluation - erectile dysfunction | 12 month post procedure
  Rate of de-novo sustained erectile dysfunction
Sexual quality of life evaluation - retrograde ejaculation | 12 month post procedure
  Rate of de-novo sustained retrograde ejaculation

CONTACTS AND LOCATIONS:
Locations (4):
- Israel (4):
  - Shamir Medical Center, Be’er Ya‘aqov
  - Bnei Zion, Haifa
  - Rabin Medical Center, Petah Tikva
  - Ziv Medical Center, Safed

IPD SHARING:
Plan to Share IPD: Undecided